CLINICAL TRIAL: NCT05244252
Title: Dexmed Vs Bupivacaine
Brief Title: Comparison of Pain ReliefofBupivacaineWith Dexmedetomidine and Bupivacaine Alone in TransversusAbdominisPlane Block For Postoperative Anelgesia in Patients Undergoing Abdominal Surgeries
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Alina Zafar, Principal investigator, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SZMC
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Pain Relief in Post Operative Patient
Keywords: Dexmeditomidine, bupivacaine, VAS, remsay sedation score
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Two groups of equal size will be included in study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Two drugs dexmeditomidine and bupivacaine will be given in TAP block
  Interventions: Drug: dexmeditomidine and bupivacaine
- Group B (Active Comparator): One drug bupivacaine will be given in TAP block
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: dexmeditomidine and bupivacaine — Transversus abdominis plane block will be given bilaterally
  Arms: Group A
Drug: Bupivacaine — bupivacaine
  Arms: Group B

SUMMARY:
Postoperative pain related to abdominal surgeries poses significant burden on the healthcare system, in terms of increased use of different analgesics, delayed ambulation, pulmonary complications, DVT, and prolonged hospital stays. Abdominal wall is major source of pain and there have been much debate in the past to bring up the effective, low cost and prolong pain relief to the patients after abdominal surgeries. But yet a consensus has to be developed about which analgesic to be used for most efficient and prolonged pain relief. Though, many studies have been done on TAP block and different combinations have been tried in TAP block, like, dexmedetomidine, midazolam, ropivacaine, but we still lack local data. Recent studies have shown very promising results in terms of efficacy and duration of block by mixing bupivacaine with dexmedetomidine, alongwith minimal side effects to the patients.

This randomised control trial will enroll 88 patients coming to Anesthesia department of Sheikh Zayed Hospital Rahim Yar Khan, for abdominal surgeries, judged on the basis of inclusion and exclusion criteria, into two groups of equal sizes. TAP block will be given to all patients bilaterally at the end of procedure after extubation in operation room. One group will be given bupivacainemixed with dexmedetomidine, while the other group will receive bupivacaine only, and they will be followed upto 12 hours postoperatively in post surgical ICU. Study protocol will be according to the ethical standards declared by Helsinki. For both the groups, HR, BP, SpO2,VAS score,rescue analgesia and sedation score stated on the clinical proforma will be assessed. After appropriate sample collection,patient data will be sorted in SPSS v23 through which statistical analysis using corresponding statistical functions and tests will be done.Quantitative data (like heart rate, mean arterial pressure, VAS score etc.) will be analysed using t-test. For qualitative variable(pain relief, bradycardia nausea etc.)chi-square test will be applied. P value </= 0.05 will be considered significant. Results of the study will be summarized and presented in final thesis.

DETAILED DESCRIPTION:
Introduction:

Pain is defined as, "an unpleasant sensory and emotional experience associated with actual or potential tissue damage or described in terms of such damage" by the international association for the study of pain. Postoperative suboptimal analgesia has very pronounced effects on the wellbeing of the patient. Patients have experienced delayed mobility, thromboembolic phenomenon, and pulmonary complications.It not only leads to prolonged stay due to delayed ambulation but also basal lung atelectasis and collapse from limited chest expansion after abdominal incision. The abdominal wall is a significant source of pain after abdominal surgery. Expected pain prevalence after hernia repair was determined as 54% and postoperative 2-year cumulative prevalence was found to be 30%.

Many methods to efficiently combat post-operative pain have been tried in the past. The multimodal approach of pain management as defined by the American Society of Anaesthesiology (ASA2012) is the administration of two or more drugs that act by different mechanisms via the same route or different route to provide optimal analgesia.Patient-controlled thoracic epidural, intravenous patient-controlled analgesia the intraperitoneal injection of local anesthetics, non-steroidal anti-inflammatory drugs, and opioids have all been part of it in different combinations.

Over the past years, the ideology of pain management has evolved from mere decreasing pain intensity to optimizing a patient's condition. The mainstay of this is to work particularly in two areas; decreasing pain scores and stress response, together with a decrease in analgesic-related side effects like nausea vomiting, and sedation. Systemic opioids have been the mainstay for postoperative analgesia for a long; but at the expense of adverse effects of nausea, vomiting, pruritus, sedation, and respiratory depression. All these issues have led to the continuous search for a better,safer, and long-lasting alternative for post-op analgesia. Though much work has been done for better understanding of the pathophysiology of postoperative pain along with the introduction of modern analgesics and delivery techniques;yet approximately 80% of the patients continue to suffer acute postoperative pain and among them, 75% experienced moderate to severe pain.

TAP block provides regional analgesia in dermatome area over T6-L1. It was initially started with the landmark technique, through lumber triangle of petit formed by external oblique muscle anteriorly, latissimussdorsi posteriorly, iliac crest inferiorly and is usually identified as a defect as 1 cam above the iliac crest in mid-axillary line. Quite several previous studies on TAP block have shown favourable results in terms of post-op pain relief, but the duration of analgesia remains an unsolved concern.Different adjuncts have been tried with bupivacaine to achieve this desired goal of long-lasting post-op analgesia with minimal side effects. Among those many studies have been done using dexamethasone,midazolam,ropivacaine, anddexmedetomidine.

Rationale:

The rationale of the study is to find out the effect of the addition of dexmedetomidine to bupivacaine on pain relief, and the demand for rescue analgesia on patients undergoing abdominal surgeries in Sheikh Zayed Hospital Rahim Yar Khan, when used in TAP block.

Past studies have shown encouraging results with the use of TAP block with or without dexmedetomidine; however, we lack local data concerning especially the patients undergoing abdominal procedures. Despite many studies performed on postoperative pain control we still have not attained gold standard criteria of multi-modal pain relief with minimal undesired effects on patients. This experimental study will pick the difference in postoperative pain relief by adding this adjunct to bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will give written informed consent
* ASA I &II
* Age between 21-45 years
* Patients undergoing abdominal surgeries
* Patients understanding VAS

Exclusion Criteria:

* Patients allergic to bupivacaine or dexmeditomidine
* Complicated procedure
* History of coagulopathy
* History of chronic use of pain medications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-04-10 (Estimated)

PRIMARY OUTCOMES:
Visual analogue score | 12 hours post operative pain will be followed
  It is a scale from 0-10 showing minimal pain on 0 and maximum pain on 10. This score is classified in to 5 categories. 0 No Pain 1-3 Mild Pain 4-6 Moderate Pain 7-9 Severe Pain 10 very severe

CONTACTS AND LOCATIONS:
Locations (1):
- Alina Zafar, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
No plans